CLINICAL TRIAL: NCT01185769
Title: Mechanism of Absorption and Distribution of Tocotrienols Under Different Food Status
Brief Title: Study of Tocotrienol Absorption and Distribution Under Different Fat Status
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: University of Malaya (Other)
Responsible Party: Wong Weng-Yew / Research Officer, Malaysian Palm Oil Board
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: PD141/09
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Last update posted 2010-08-20 (Estimated); Status verified 2010-08

CONDITIONS: Absorption
Keywords: Vitamin E; Absorption
MeSH Terms: interventions — Tocotrienols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- High fat (Experimental): 500 mg of tocotrienol will be administered at single dose after consumption of high fat diet
  Interventions: Dietary Supplement: Tocotrienol
- Low fat (Experimental): 500 mg of tocotrienol will be administered at single dose after consumption of low fat diet
  Interventions: Dietary Supplement: Tocotrienol

INTERVENTIONS:
Dietary Supplement: Tocotrienol — 500 mg of tocotrienol will be administered after consumption of high fat diet
  Arms: High fat
Dietary Supplement: Tocotrienol — 500 mg of tocotrienol will be administered after consumption of low fat diet
  Arms: Low fat

SUMMARY:
Despite the emerging interest in tocotrienols, the absorption of tocotrienols in humans remains unclear especially with different fat diets.This study aimed at evaluating the absorption and distribution of tocotrienols in plasma and lipoproteins in associations with high and low fat diets. Different fat level will affect the absorption and distribution of tocotrienols

DETAILED DESCRIPTION:
There is a possibility that the absorption and distribution of tocotrienols may occur differently compared with tocopherols, especially under different fat status

ELIGIBILITY:
Inclusion Criteria:

* male aged 22-25
* body mass index 18.5 < X < 30 kg/m2
* plasma cholesterol < 5.2 mmol/L,
* TAG < 1.7 mmol/L

Exclusion Criteria:

* history of cardiovascular disease
* diabetic
* body mass index < 18.5 or > 30 kg/m2
* plasma cholesterol > 5.2 mmol/L,
* TAG > 1.7 mmol/L
* hypertension
* currently taking Vitamin E supplement
* current use of medication
* smoking.

Ages: 22 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2009-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Difference in absorption and distribution of Tocoterienols during high fat and low fat meal by measuring the plasma, chylomicron, and HDL level of tocotrienol | 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 24 hours after tocotrienol administration and in take of designated meal

CONTACTS AND LOCATIONS:
Overall Officials: Weng-Yew Wong, Bsc, Principal Investigator — Malaysia Palm Oil Board
Locations (1):
- Malaysian Palm Oil Board, Bangi, Selangor, Malaysia